CLINICAL TRIAL: NCT01839032
Title: A Phase II Study of Cisplatin With Intravenous and Oral Vinorelbine as Induction Chemotherapy Followed by Concomitant Chemotherapy With Oral Vinorelbine and Cisplatine for Locally Advances Non-small Cell Lung Cancer
Brief Title: Oral Vinorelbine as Induction Chemotherapy Followed Concomitant Chemoradiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 041316
Record Dates: First submitted 2013-04-05; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vinorelbine cisplatin radiotherapy (Experimental): Induction period + radio chemotherapy
  Interventions: Drug: Vinorelbine cisplatin radiotherapy

INTERVENTIONS:
Drug: Vinorelbine cisplatin radiotherapy — During the induction period, patients received chemotherapy for two 3-week cycles. Bolus intravenous vinorelbine 25 mg/m², was administered on day 1, then cisplatin 80 mg/m² was administered over 1-hour infusion. Vinorelbine 60 mg/m² was also administered on day 8.
  Patients with objective response (OR) or no change (NC) continued the concomitant period (CP) including two additional 3-week cycles of radio chemotherapy (vinorelvine 20 mg D1 D3 D5 Cisplatin 80 mg/m² 66 Gy).
  Other Names: Navelbine

SUMMARY:
Patients (pts) with stage IIIA/IIIB NSCLC received NVBiv 25 mg/m² + CDDP 80 mg/m² on D1 and NVBo 60 mg/m² on D8 every 3 weeks (q3w) for 2 cycles as induction. Pts with response or non change received NVBo 20 mg fixed dose on D1 D3 D5 + CDDP 80 mg/m² on D1 q3w for 2 more cycles during RT(66 Gy/6.5 w).

DETAILED DESCRIPTION:
Vinorelbine (NVB) + CDDP is considered a standard trt in induction or concomitantly with RT (Vokes, Fournel, Krzakowski). NVBo simplifies the administration of trt and provides the same efficacy as intravenous NVB (NVBiv). In order to assess this and to improve the tolerance, a trial was started with NVBiv and NVBo + CDDP as induction followed by a fractionated administration of NVBo + CDDP during RT.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed stage IIIA (only N2),
* dry IIIB previously untreated inoperable NSCLC,
* 18 to 75 years old,
* Karnofsky Performance Status (KPS) ≥ 80%,
* weight loss ≤ 10% within the previous 3 months,
* normal organ functions were eligible.
* at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST version 1.0) [10].

Exclusion Criteria:

* stages I, II, IIIA (excepted N2), IIIB with pleural effucion and stage IV,
* pregnant or breastfeeding women. Women of Childbearing Age: Women of childbearing potential should take reliable contraceptive measures
* Symptomatic Neuropathy > grade 1,
* associated Pathology and/or not controled diseases(cardiac insuficiency, myocardial infarction within 3 months before the inclusion ; hypertension, arythmia or uncontroled hypercalcémia; infection requiering iv antibiotic administration within 2 weeks before inculion),
* other associated cancer with the exception of cervical carcinoma in situ or skin cancer baso-cellular correctely treated,
* Previous treatment with an other antineoplasic,
* Known hypersensibility to drugs with a similar chemical structure ti this studied.
* important malabsorbtion syndrom or disease of gastro-intestinal track,
* Participation to another clinical trial within 30 days before inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Disease controle | up to 3 years

SECONDARY OUTCOMES:
- duration of response (DR) | up to 3 years
  Secondary endpoints were duration of response (DR), progression-free survival (PFS), and overall survival (OS), calculated by the Kaplan-Meier method. The safety analysis reported the worst grade of the adverse events (NCI CTC v. 2.0) for the safety population.

OTHER OUTCOMES:
- progression-free survival (PFS) | up to 3 years
- overall survival (OS), | up to 3 years
- safety | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Zalcmann, professor, Study Chair — Baclesse, Caen, France
Locations (1):
- CHU CAEN, Caen, France

REFERENCES:
- [Derived] Lerouge D, Riviere A, Dansin E, Chouaid C, Dujon C, Schott R, Lavole A, Le Pennec V, Fabre E, Crequit J, Martin F, Dehette S, Fournel P, Precheur-Agulhon B, Lartigau E, Zalcman G. A phase II study of cisplatin with intravenous and oral vinorelbine as induction chemotherapy followed by concomitant chemoradiotherapy with oral vinorelbine and cisplatin for locally advanced non-small cell lung cancer. BMC Cancer. 2014 Mar 30;14:231. doi: 10.1186/1471-2407-14-231. PMID 24678902